CLINICAL TRIAL: NCT02941718
Title: Examination of Sleep, Smoking Cessation, and Cardiovascular Health
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Freda Patterson, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 887213
Record Dates: First submitted 2016-08-16; First posted 2016-10-21 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Nicotine Dependence
Keywords: Smoking; Smoking cessation; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (2):
- Sleep Advancement Counseling (Experimental): Participants will receive a 15-week intervention targeting smoking cessation and sleep counseling intervention.
  Smoking Cessation intervention components include:
  * 6 individual smoking cessation sessions over 15 weeks (week 1, 3, 4, 7, 11, 15)
  * 12 weeks of the quit-smoking drug chantix. The standard dosing will be used - 0.5 mg once per day for days 1-3, 0.5my twice per day for days 4-7; and 1mg twice per day from week 3 until the end of treatment.
  Sleep counseling components in the form of CBT for insomnia will be given as part of the smoking cessation counseling.
  Interventions: Behavioral: Sleep Advancement Counseling
- General Health Intervention (Active Comparator): Participants will receive a 15-week intervention targeting smoking cessation and general health information.
  Smoking Cessation intervention components include:
  * 6 individual smoking cessation sessions over 15 weeks (week 1, 3, 4, 7, 11, 15)
  * 12 weeks of the quit-smoking drug chantix. The standard dosing will be used - 0.5 mg once per day for days 1-3, 0.5my twice per day for days 4-7; and 1mg twice per day from week 3 until the end of treatment.
  The general health information counseling will be given as part of the smoking cessation counseling and topics include diet, physical activity, oral health, cancer screening and skin protection.
  Interventions: Behavioral: General Health Information

INTERVENTIONS:
Behavioral: Sleep Advancement Counseling — Participants will receive cognitive behavioral counseling on achieving adequate sleep duration.
  Arms: Sleep Advancement Counseling
Behavioral: General Health Information — Participants will receive educational information on general health topics including diet, physical activity, skin protection, oral health and cancer screenings.
  Arms: General Health Intervention

SUMMARY:
Most treatment-seeking smokers will fail in their attempts to quit smoking in the early days and weeks of quitting. Poor sleep (e.g., short duration) is an overlooked, but important nicotine withdrawal symptom that can affect up to 80% of treatment seeking smokers and predicts relapse. Addressing sleep deficits could promote cessation, particularly in smokers who may be vulnerable to poor sleep in one or more sleep metrics even before quitting. This study will address this conceptual and empirical gap by conducting a 15-week proof-of-concept study to determine whether standard smoking cessation treatment can be optimized with a multi-metric sleep advancement counseling intervention.

DETAILED DESCRIPTION:
The current study is a randomized controlled trial designed to test the impact and efficacy of a sleep advancement counseling (SAC) protocol in response to standard nicotine dependence treatment (behavioral counseling + varenicline) in a sample of 90 treatment seeking smokers from the greater Newark city/Newcastle county area. Following eligibility assessment, which include an overnight polysomnography (sleep study), 90 eligible and consenting treatment-seeking smokers will be randomized to either the experimental smoking cessation + SAC (N=60), or the control, smoking cessation + general health education (GHE) alone (N=30) condition. Participants will complete six in-person counseling sessions over a 15-week treatment period (wks 1, 3, 4,7,11,15) As part of the smoking cessation treatment protocol, eligible participants will receive 12 weeks of FDA-approved smoking cessation medication, Varenicline, during week 3-15. An end of treatment (week 15) and a 12-week follow-up (week 27) assessment will be conducted in-person to allow for the objective assessment of smoking status and cardiovascular markers.

ELIGIBILITY:
Inclusion Criteria:

1. adults (>18 -65) who smoke at least 8 cigarettes/day;
2. Report wanting to quit smoking in the next month
3. No current diagnosis of psychosis or bipolar disorder.
4. able to communicate in English and provide written informed consent for study procedures
5. able to use varenicline safely.
6. No current diagnosis of any sleep disorders (except of insomnia)
7. Have access to a smart phone or tablet own the home

Exclusion Criteria:

1. Current enrollment or plans to enroll in another smoking cessation program and/or use a nicotine substitute (e.g., e-cigarettes) in the next 6 months,
2. Current use of illicit drugs (e.g., cocaine, opioids, or methamphetamines),
3. Current alcohol consumption that exceeds 14 standard alcoholic drinks/week for men, and more than 7 for women.
4. Current use or recent discontinuation (within last 14 days) of anti-psychotic and/or bipolar disorder medications,
5. Women who are pregnant, planning a pregnancy within the next 6 months, or lactating,
6. Uncontrolled hypertension (SBP >160 or DBP >100)
7. Current sleep disorder or use of sleep medication
8. History of heart disease, stroke or MI, unstable angina, abnormal heart rhythms, or tachycardia (if stable, requires Study Physician approval),
9. Any current suicidal ideation, or self-reported suicide attempt
10. Current or past diagnosis of psychotic or bipolar disorder
11. Currently working night/rotating shift.
12. Allergy to Varenicline
13. Unstable or untreated moderate or severe depression as assessed by the center for epidemiology studies depression scale 16 for higher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Carbon Monoxide Level | 15-week
  % of participants with a CO level of 10 or fewer parts per million (ppm)

SECONDARY OUTCOMES:
Objective Sleep Duration and Timing | 15-weeks
  Will be measured using a motion-logger accelerometer device. Participants will wear the lotion logger watches on their non-dominant wrist at key points during the study (weeks 1, 4, 15). Data will be collected at 1min epochs.

CONTACTS AND LOCATIONS:
Overall Officials: Freda Patterson, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patterson F, Malone SK, Lozano A, Grandner MA, Hanlon AL. Smoking, Screen-Based Sedentary Behavior, and Diet Associated with Habitual Sleep Duration and Chronotype: Data from the UK Biobank. Ann Behav Med. 2016 Oct;50(5):715-726. doi: 10.1007/s12160-016-9797-5. PMID 27056396
- [Background] Malone SK, Patterson F, Lu Y, Lozano A, Hanlon A. Ethnic differences in sleep duration and morning-evening type in a population sample. Chronobiol Int. 2016;33(1):10-21. doi: 10.3109/07420528.2015.1107729. Epub 2015 Dec 10. PMID 26654569
- [Background] Patterson F, Jepson C, Loughead J, Perkins K, Strasser AA, Siegel S, Frey J, Gur R, Lerman C. Working memory deficits predict short-term smoking resumption following brief abstinence. Drug Alcohol Depend. 2010 Jan 1;106(1):61-4. doi: 10.1016/j.drugalcdep.2009.07.020. Epub 2009 Sep 5. PMID 19733449
- [Background] Patterson F, Jepson C, Strasser AA, Loughead J, Perkins KA, Gur RC, Frey JM, Siegel S, Lerman C. Varenicline improves mood and cognition during smoking abstinence. Biol Psychiatry. 2009 Jan 15;65(2):144-9. doi: 10.1016/j.biopsych.2008.08.028. Epub 2008 Oct 8. PMID 18842256
- [Background] Patterson F, Kerrin K, Wileyto EP, Lerman C. Increase in anger symptoms after smoking cessation predicts relapse. Drug Alcohol Depend. 2008 May 1;95(1-2):173-6. doi: 10.1016/j.drugalcdep.2008.01.013. Epub 2008 Mar 6. PMID 18328642

DOCUMENTS (1):
  • Informed Consent Form (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02941718/ICF_000.pdf